CLINICAL TRIAL: NCT05664087
Title: Effect of Photodynamic Therapy on Soft Tissue Healing After Tooth Extraction at Sites of Periodontal Infection: a Randomized Controlled Clinical Trial
Brief Title: Effect of Photodynamic Therapy on Soft Tissue Healing After Tooth Extraction at Sites of Periodontal Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Dental Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Peihui Ding, Principal Investigator, The Dental Hospital of Zhejiang University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DHZhejiangU-2022(197)
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Debridement of tooth extraction sockets was assisted by photodynamic equipment
  Interventions: Drug: Dental diode laser device Paiwei™（Zhengzhou Gata biotechnology Co.,Ltd.,China） which was 650-670nm with a power of 160mw-220mw.
- control group (No Intervention): Routine tooth extraction and debridement were performed

INTERVENTIONS:
Drug: Dental diode laser device Paiwei™（Zhengzhou Gata biotechnology Co.,Ltd.,China） which was 650-670nm with a power of 160mw-220mw. — The tooth extraction sockets were filled with photosensitizer methylene blue. The guide head of the laser periodontal therapy instrument (Dental diode laser device Paiwei™（Zhengzhou Gata biotechnology Co.,Ltd.,China） which was 650-670nm with a power of 160mw-220mw.) was placed in the tooth extraction sockets to probe and move around the tooth extraction sockets for 1 minute. At the end of irradiation, a cotton ball dipped in saline was used to wipe the guide head and rinse the photosensitizer out of the socket
  Other Names: The disposable dental Treatment Kits Paiwei™（Zhengzhou Gata biotechnology Co.,Ltd.,China）
  Arms: Experimental group

SUMMARY:
Main Purpose: To evaluate the effect of photodynamic therapy on soft tissue healing after tooth extraction at periodontal infection site, and to compare the effect on pain degree and bone tissue remodeling after tooth extraction.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of photodynamic therapy (PDT) on soft tissue healing and bone remodeling in tooth extraction sockets after tooth extraction. The enrolled patients will be randomized into two groups. The control group used conventional tooth extraction to clean the wound, and the experimental group used photodynamic therapy to help clean the wound. Seven days and 14 days after extraction, the area of extraction socket was measured, the healing rate of extraction socket was calculated, and Landry, Turnbull and Howley soft tissue healing index was measured. The degree of pain was recorded at 6h, 1 day, 2 days and 3 days after tooth extraction. Bone remodeling indexes were measured at 1 month after tooth extraction.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 18 to 65 years old;
* Patients with extensive periodontitis of the whole mouth;
* There was a deep periodontal pocket with PD≥5mm and at least one adjacent tooth at the extraction site;
* Periodontitis was controlled, and the extraction site and adjacent teeth were not in the acute inflammation or infection stage;
* The extraction site has a hopeless prognosis or no preservation value, and it is the first and second molars or maxillary wisdom teeth that erupt in a positive position

Exclusion Criteria:

* pregnant and lactating women;
* patients with systemic diseases that may affect the ability of postoperative healing (such as patients with radiotherapy and chemotherapy, history of hematological diseases, and uncontrolled disease) Diabetes mellitus, etc.);
* long-term use of drugs known to affect bone metabolism or mucosal healing such as bisphosphonates and non-steroidal anti-inflammatory drugs;
* smoking > 10 cigarettes per day;
* root breakage or gingival tear occurred during tooth extraction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Wound healing rate at 7 days | baseline;at 7 days
  （The size of the tooth extraction wound area at 7 days）/(The size of the tooth extraction wound area at baseline)

SECONDARY OUTCOMES:
Landry, Turnbull and Howley soft tissue healing index | baseline, at 7 days; at 14days
  Soft tissue index of healing wound after tooth extraction
Degree of pain | at 6 hours; at 1 day; at 2 days; at 3 days
  VAS score was used to evaluate the pain degree of tooth extraction trauma. A score of 0 indicates no pain and a score of 10 indicates severe pain.
Changes in Bone Mineral density | baseline, at 1 month
  Changes in Bone Mineral density
Bone height changes | baseline, at 1 month
  Bone height changes
Wound healing rate at 14 days | baseline;at 14 days
  （The size of the tooth extraction wound area at 14 days）/(The size of the tooth extraction wound area at baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Peihui Ding, Doctor, Principal Investigator — The Affiliated Stomatology Hospital of Zhejiang University School of Medicine
Locations (1):
- The Affiliated Stomatology Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No